CLINICAL TRIAL: NCT00056225
Title: High Dose Supplements to Reduce Homocysteine and Slow the Rate of Cognitive Decline in Alzheimer's Disease (Vitamins to Slow Alzheimer's - VITAL)
Brief Title: VITAL - VITamins to Slow ALzheimer's Disease (Homocysteine Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: Alzheimer's Disease Cooperative Study (ADCS) (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IA0041
Record Dates: First submitted 2003-03-07; First posted 2003-03-10 (Estimated); Last update posted 2009-06-12 (Estimated); Status verified 2009-06

CONDITIONS: Alzheimer's Disease
Keywords: homocysteine
MeSH Terms: conditions — Alzheimer Disease | interventions — Folic Acid; Vitamin B 6; Vitamin B 12

INTERVENTIONS:
Drug: Folate
Drug: Vitamin B6
Drug: Vitamin B12

SUMMARY:
The purpose of this study is to determine whether reduction of homocysteine levels with high-dose folate (folic acid), B6, and B12 supplementation will slow the rate of cognitive decline in persons with Alzheimer's disease.

DETAILED DESCRIPTION:
Blood levels of homocysteine are elevated in Alzheimer's disease (AD), and hyperhomocysteinemia may contribute to disease pathophysiology by vascular and direct neurotoxic mechanisms. Homocysteine levels can be reduced by administration of high dose supplements of folate (folic acid) and vitamins B6 and B12. The proposed study is for a multicenter, randomized, controlled clinical trial to determine whether reduction of homocysteine levels with high-dose folate/B6/B12 supplementation will slow the rate of cognitive decline in subjects with AD.

This will be a parallel design study, including two groups of unequal size: 60% of subjects will receive daily high-dose supplements (folate 5mg, vitamin B6 25mg, vitamin B12 1 mg), and 40% will receive an identical looking placebo. The duration of treatment will be 18 months, and participants will make eight visits to the assigned study site for safety and efficacy assessments of the medications. The primary outcome measure will be the longitudinal decline in the ADAScog, a psychometric instrument that evaluates memory, attention, reasoning, language, orientation and praxis (Rosen et al 1984). To power the trial to detect a 25% reduction in rate of ADAScog decline (80% power, alpha=0.05, drop-out estimate 20%, drop-in estimate 10%), it will enroll a total of 400 participants. Persons of minority racial groups are also being recruited, although all participants must be able to speak either English or Spanish.

ELIGIBILITY:
Inclusion Criteria:

* National Institute of Neurological Disorders and Stroke (NINDS)/Alzheimer's Disease and Related Disorders Association (ADRDA) criteria for probable Alzheimer's disease.
* Mini-Mental Status Examination (MMSE) score between 14 and 26, inclusive
* Stable medical condition for 3 months
* Stable medications for 4 weeks prior to the screening visit
* Physically acceptable for this study as confirmed by medical history, physical exam, neurologic exam and clinical laboratory tests
* Supervision available for administration of study medications
* Study partner to accompany subject to all scheduled visits
* Fluent in English or Spanish
* Modified Hachinski equal to or less than 4 CT or magnetic resonance imaging (MRI) since onset of memory impairment demonstrating absence of clinically significant focal lesion
* Able to complete baseline assessments
* 6 years of education or work history sufficient to exclude mental retardation
* Able to ingest oral medication

Exclusion Criteria:

* B12 or folate deficiency
* Renal insufficiency (serum creatinine >=2.0)
* Active neoplastic disease (skin tumors other than melanoma are not exclusionary; patients with stable prostate cancer may be included at the discretion of the project director)
* Use of another investigational agent within 2 months
* History of clinically significant stroke
* Current evidence or history in the past 2 years of epilepsy, focal brain lesion, head injury with loss of consciousness and/or immediate confusion after the injury, or DSM-IV criteria for any major psychiatric disorder including psychosis, major depression, bipolar disorder, alcohol or substance abuse
* Blindness, deafness, language difficulties or any other disability which may prevent the subject from participating or cooperating in the protocol

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2003-01; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Aisen, MD, Principal Investigator — Georgetown University, Department of Neurology
Locations (38):
- United States (38):
  - University of Alabama, Birmingham, Alabama
  - Mayo Clinic, Scottsdale, Scottsdale, Arizona
  - Sun Health Research Institute, Sun City, Arizona
  - University of Arizona, Arizona Health Sciences Center, Tucson, Arizona
  - University of California, Irvine, Institute for Brain Aging and Dementia, Irvine, California
  - University of California, San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California, Davis, Sacramento, California
  - Yale University, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - Howard University, Washington D.C., District of Columbia
  - Mayo Clinic, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush Presbyterian/St. Lukes Medical Center, Rush Alzheimer's Disease Center, Chicago, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Indiana University, Indianapolis, Indiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Nevada School of Medicine, Center for Cognitive Aging, Las Vegas, Nevada
  - ClinSearch, Kenilworth, New Jersey
  - New York University Medical Center, New York, New York
  - Mt. Sinai School of Medicine, New York, New York
  - Columbia University, New York, New York
  - University of Rochester Medical Center, Alzheimer's Disease Center, Rochester, New York
  - University Memory and Aging Center, Case Western Reserve University/University Hospitals of Cleveland, Cleveland, Ohio
  - Oregon Health and Science University, Oregon Aging and Alzheimer's Disease Center, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Memorial Hospital of Rhode Island, Alzheimer's Disease and Memory Disorder Clinic, Pawtucket, Rhode Island
  - Medical University of South Carolina, North Charleston, South Carolina
  - University of Texas, Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Seshadri S, Beiser A, Selhub J, Jacques PF, Rosenberg IH, D'Agostino RB, Wilson PW, Wolf PA. Plasma homocysteine as a risk factor for dementia and Alzheimer's disease. N Engl J Med. 2002 Feb 14;346(7):476-83. doi: 10.1056/NEJMoa011613. PMID 11844848
- [Background] Aisen PS, Egelko S, Andrews H, Diaz-Arrastia R, Weiner M, DeCarli C, Jagust W, Miller JW, Green R, Bell K, Sano M. A pilot study of vitamins to lower plasma homocysteine levels in Alzheimer disease. Am J Geriatr Psychiatry. 2003 Mar-Apr;11(2):246-9. PMID 12611755
- [Background] Kruman II, Kumaravel TS, Lohani A, Pedersen WA, Cutler RG, Kruman Y, Haughey N, Lee J, Evans M, Mattson MP. Folic acid deficiency and homocysteine impair DNA repair in hippocampal neurons and sensitize them to amyloid toxicity in experimental models of Alzheimer's disease. J Neurosci. 2002 Mar 1;22(5):1752-62. doi: 10.1523/JNEUROSCI.22-05-01752.2002. PMID 11880504
- [Result] Aisen PS, Schneider LS, Sano M, Diaz-Arrastia R, van Dyck CH, Weiner MF, Bottiglieri T, Jin S, Stokes KT, Thomas RG, Thal LJ; Alzheimer Disease Cooperative Study. High-dose B vitamin supplementation and cognitive decline in Alzheimer disease: a randomized controlled trial. JAMA. 2008 Oct 15;300(15):1774-83. doi: 10.1001/jama.300.15.1774. PMID 18854539